CLINICAL TRIAL: NCT00944086
Title: A Prospective Randomized Clinical Study:Oxygen Concentration Should be Kept at the Lowest Possible Level During Recruitment Manoeuvres
Brief Title: Oxygen Concentration Should be Kept at the Lowest Possible Level During Recruitment
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Other Study IDs: Akaratas
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Laparoscopic Surgery
Keywords: Recruitment; Oxygen Concentration; pneumoperitoneum; laparoscopy
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Recruitment Manoeuvre ,Laparoscopy
  Interventions: Other: Recruitment Manoeuvre

INTERVENTIONS:
Other: Recruitment Manoeuvre — Recruitment Manoeuvre

SUMMARY:
In This Study, Our Goal is to Compare the Effects of Recruitment Manoeuvre Which is Applied With Different Oxygen Concentrations on Oxygenation and Respiratory Mechanics During Pneumoperitoneum

DETAILED DESCRIPTION:
Detailed Description:

"Recruitment manoeuvre" which has been defined and become popular in the recent years is nowadays widely accepted and applied. The positive effects of the recruitment manoeuvre during and after surgery on respiratory mechanics and oxygenation have been reported. The duration and the applied pressure values of recruitment manoeuvre have been defined well and in detail regarding the definitions for this manoeuvre (1-3). Despite these definitions, no detailed information has been provided on the effects of the oxygen and oxygen concentration during recruitment manoeuvre .

Atelectasis develops after the induction of anaesthesia, even in healthy subjects, and is associated with an increase in intraoperative shunt leading to impairment of gas exchange (4). It is well known that in patients, who have undergone mechanical ventilation with high oxygen concentration levels, oxygen replaces the less insoluble nitrogen. Partial oxygen pressure increases with the implementation of oxygen in high concentrations, and the oxygen flow into the blood increases. But when the gas flow into the blood is more than inspired, absorption atelectasis develops in lungs - due to appliance of high oxygen concentration. Atelectasis may also develop due to different reasons such as failure in secretion clearance during the surgery, replacement of nitrogen with inhalation anaesthetics and appliance of pneumoperitoneum.

In the recent years, many studies have analyzed the effects of recruitment manoeuvre during pneumoperitoneum and laparoscopic surgery on respiratory mechanics and oxygenation, and reported the benefits of recruitment in these operations (4-6).

In this study, our goal is to compare the effects of recruitment manoeuvre which is applied with different oxygen concentrations on oxygenation and respiratory mechanics during pneumoperitoneum.

ELIGIBILITY:
Exclusion Criteria:

* Patients, who were older than 65 years,
* had respiratory system and cardiovascular diseases,
* used medication that could affect the respiratory function or smokers have been excluded.

Ages: 27 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study has been applied on 32 cases which have undergone laparoscopic cholecystectomy.
Sampling Method: Probability Sample
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cerrahpasa School of Medicine, Istanbul, Turkey (Türkiye)